CLINICAL TRIAL: NCT03520855
Title: Contribution of a Serious Game in the Therapeutic Education of Type 1 Diabetes Paediatric Patients
Brief Title: Serious Game in the Therapeutic Education of Type 1 Diabetes Paediatric Patients
Acronym: eDIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K150907J; 2017-A02052-51 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-04-27; First posted 2018-05-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Paediatrics patients
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ETP + Serious game (Experimental): patients receiving the serious game additionally to the classic therapeutic education
  Interventions: Other: Serious game; Behavioral: ETP
- ETP (Active Comparator): patients under classic therapeutic education
  Interventions: Behavioral: ETP

INTERVENTIONS:
Other: Serious game — DIVE software will be accessible via internet, children and parents will have to their disposition a room at the hospital specifically to work on the software. The DIVE software is organized in chapters, each matches an item of the therapeutic education process and ends with a knowledge assessment. The child has to end every chapter and succeed every evaluation to pursue on the next chapter. Measures will be taken in order to avoid contamination bias between groups. Children will have to connect to DIVE 2 times per week for a time duration of at last 1 hour.
  Arms: ETP + Serious game
Behavioral: ETP — Initial therapeutic education only will be applied in this group, with the help of doctors and nurses, based on theoretical educational lessons, reported on the AJD book.
  Health education sessions will also be taught by nurses.

SUMMARY:
The aim of this study is to evaluate the contribution of a serious game in the reinforcement of knowledge acquired during therapeutic education of type 1 diabetes paediatric patients.

This evaluation will take place within 3 months of the diagnosis.

DETAILED DESCRIPTION:
Type 1 diabetes gather multiple metabolic pathologies secondary to a deficiency in insulin secretion or insulin action, characterized by chronic hyperglycaemia. Diagnosis is based on fasting glycaemia above 1.26 g/l or above 2 g/l any time of the day.

Currently, it is recommend initial therapeutic education additionally to insulin therapy, in the type 1 diabetes care. Initial therapeutic education's role is to develop 3 specific skills : self-care skills, safety skills and adaptation skills. This approach gives to the patient the abilities to monitor himself, to handle emergency situations and to modify his lifestyle to treat his disease correctly.

In the serious game, the patient will directly evolve in a virtual environment, with places reflecting his real life such as paediatric diabetology centre, hospital, home, school. He will have to complete quests with his own virtual avatar, that reflect situations his disease can confront him to. Each quest ends with a questionnaire.

The principal objective of this research is to evaluation the contribution of a serious game (DIVE) in the reinforcement of knowledge acquired during therapeutic education of type 1 diabetes paediatric patients.

This research is designed in two arms, gathering 100 patients, each arm has 50 patients. Both arms benefit initial therapeutic education, except the experimental group which is added a serious game .

To measure the impact of the serious game,investigators will compare HbA1c dosage between groups (with HPLC technique), 3 months after diagnosis; but also the number of hypo or hyperglycaemia in the month before M3 final consultation. They will also evaluate self-care skills and safety skills with role-plays at the end of hospitalisation and 3 months later. Technical gestures will also be evaluated by referent nurses.

Evaluation of the patient's well-being will take place with two types of questionnaire, WHO-Five and DOQLY during M3 final consultation.

This research will bring essential information on the development of video games in other paediatric chronic diseases, as a first step in the development of the use of video games in therapeutic care of type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Child aged from 10 to 17 and 8 months
* Child with a type 1 diabetes (inclusion within 96 hours following the diagnosis, except for patients admitted to intensive care for whom an additional 48-hour period is accepted for their inclusion). Diagnosis will be confirmed based on one of the classic diagnostic criteria: venous glycaemia above 2 g / l, presence of polyuropolydipsic syndrome, presence of weight loss, presence of ketonuria (equivalent to at least one cross in urine or> 0.5mmol / l in blood)
* Child with internet access and with a computer or a tablet or a mobile phone in at least one of the two parents or legal representative(s)
* Informed consent signed by parents or legal representative(s) (only one parent possible)
* Beneficiary of a social security system

Exclusion Criteria:

* No internet access or no computer or no tablet or no mobile phone at home available
* No French language proficiency of the infant or legal representative(s)
* Inability to understand the game's instructions
* Inability to understand or fill the consent

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Diapason questionnaire (Aide aux Jeunes Diabètes) | 3 months
  50 questions (disease, treatment, food,…)

SECONDARY OUTCOMES:
HbA1c dosage | 3 months
  Glycemia follow-up with a self-monitoring book in each arm
Number of hypo or hyperglycaemia | 3 months
  Statement of the number of hypo or hyperglycaemia within the months preceding the consultation
Evaluation of self-care skills | 3 months
  Evaluation of self-care skills with role-plays and assessment of feelings of competence from their DT1 (scorecard, Barrow chart )
Evaluation of well-being with WHOFIVE | 3 months
  Evaluation of patient's well-being with auto-questionnaires
Evaluation of well-being with DQOLY | 3 months
  Evaluation of patient's well-being with auto-questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jacques BELTRAND, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No